CLINICAL TRIAL: NCT01613924
Title: Efficacy of a Handheld Heat Based Device for the Spot Treatment of Mild to Moderate Acne Vulgaris: A Controlled Study to Determine Time to Resolution of Individual Inflammatory Lesions Using an Over-the-counter Acne Heat Device.
Brief Title: Efficacy of Handheld Acne Heat Device
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding and resources
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12-00792
Record Dates: First submitted 2012-05-30; First posted 2012-06-07 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heat based treatment/no treatment (Placebo Comparator): Split face treatment with handheld acne heat based device and no treatment
  Interventions: Device: Split face: handheld acne heat based device (Zeno Hot Spot) and no treatment
- Heat based treatment/benzoyl peroxide (Active Comparator): Split face treatment with handheld acne heat based device and benzoyl peroxide 4%
  Interventions: Device: Split face: handheld acne heat based device, Zeno Hot Spot, and topical benzoyl peroxide 4%

INTERVENTIONS:
Device: Split face: handheld acne heat based device (Zeno Hot Spot) and no treatment — Subjects will apply the actual device to every inflammatory acne facial lesion on one half of the face and no treatment to every inflammatory acne lesion on the other half of the face at 6 hour intervals for a total of 3 treatments. Follow up will occur daily over a 5 day period.
  Arms: Heat based treatment/no treatment
Device: Split face: handheld acne heat based device, Zeno Hot Spot, and topical benzoyl peroxide 4% — Subjects will apply the actual device to every inflammatory acne facial lesion on one half of the face at 6 hour intervals for a total of 3 treatments. Subjects will apply benzoyl peroxide to the other half of the face daily for 5 days.
  Arms: Heat based treatment/benzoyl peroxide

SUMMARY:
The aim of our study is to determine the time to resolution of individual acne lesions using a popular handheld heat based device in comparison to no treatment and to standard topical therapy with benzoyl peroxide in order to determine its effectiveness in the spot treatment of acne vulgaris. Patient satisfaction and potential side effects will be examined as well.

ELIGIBILITY:
Inclusion Criteria:

* Are 12- 64 years old
* Have an Investigator's Global Assessment of greater than or equal to 2
* Have 8-16 inflammatory acne facial lesions (papules and pustules)

Exclusion Criteria:

* Have any severe facial acne at baseline, including large acne lesions and cysts (nodulocystic acne)
* Have used any topical anti-acne medications, systemic antibiotics, and/or systemic corticosteroids 4 weeks before the study start
* Have used oral acne medications, such as Accutane (systemic retinoid), 6 months before the study start
* Have had a facial procedure 2 weeks before the study start
* Are nursing or pregnant
* Are using any oral contraceptives that have a specific anti-androgenic action or if you have started using a new oral contraceptive 12 weeks before the study start
* Are using any medications known to exacerbate acne
* Have a known hypersensitivity or allergy to benzoyl peroxide or any of the vehicle constituents
* Have a beard or facial hair that could interfere with study evaluations

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Time to resolution of individual acne lesions | 5 days
  Subjects will be photographed daily and the progression of individual acne lesions will be followed. Time to resolution of each lesion will be determined for the various treatment groups.

SECONDARY OUTCOMES:
Device tolerability | 5 days
  Device tolerability will be assessed daily by asking the subject about adverse effects experienced from the treatments. At the end of 5 days, subjects will be asked to rate the various treatments based on ease of use and how much the side effects bothered him or her.
Split-face investigator's static global assessment | 5 days
  Split-face investigator's static global assessments will be conduced daily on subjects for 5 days.
Acne lesion counts | 5 days
  Lesion counts will be performed daily for 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Humphrey, MD, FRCPC, Principal Investigator — UBC Department of Dermatology and Skin Science
Locations (1):
- Skin Care Centre, Vancouver, British Columbia, Canada